CLINICAL TRIAL: NCT01775982
Title: Validation of a French Version of the Confusion Assessment Method (CAM): a Diagnostic Tool for Acute Confusion Among the Elderly
Brief Title: Validation of a French Version of the Confusion Assessment Method (CAM)
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: PHRC-N/2011/VA-04; 2011-A01161-40 (Other: ANSM)
Record Dates: First submitted 2013-01-23; First posted 2013-01-25 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2017-01

CONDITIONS: Confusion; Delirium
Keywords: French language validation; The Confusion Assessment Method (CAM)
MeSH Terms: conditions — Confusion; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study population: See inclusion and exclusion criteria.
  Intervention: Psychiatric evaluation Intervention: Geriatric evaluation
  A potential intervention order effect will be taken into account by balancing in each center the number of evaluations beginning with the geriatric assessment and those starting with the psychiatric assessment.
  Interventions: Other: Psychiatric evaluation; Other: Geriatric evaluation

INTERVENTIONS:
Other: Psychiatric evaluation — This evaluation is carried out in several stages:
  * Assessment of cognitive functioning;
  * Interview with a relative;
  * Interview with caregivers;
  * Evaluation of the presence of delirium according to DSM-IV criteria;
  * Evaluation of the presence of anxiety, depressive syndrome, dementia or other DSM IV;
  * Reports of adverse events.
  A potential intervention order effect will be taken into account by balancing in each center the number of evaluations beginning with the geriatric assessment and those starting with the psychiatric assessment.
Other: Geriatric evaluation — This evaluation includes a brief interview with a caregiver, diverse scorings (CAM, Delirium Index, Mini Geriatric Depression Scale, Modified Early Warning Score, Clinical Global Impression sclae, Algo Plus), and adverse event reporting.
  CAM scoring is carried out by a trained geriatrician and a trained nurse and/or a psychologist.
  A potential intervention order effect will be taken into account by balancing in each center the number of evaluations beginning with the geriatric assessment and those starting with the psychiatric assessment.

SUMMARY:
To validate the French version of the CAM, a multicenter diagnostic study will be conducted. The principle of this study is identical to the study of Inouye which initially validated the CAM in 1990. This is to verify the diagnostic properties of the CAM (French version) compared to the gold standard represented by the confused state of psychiatric diagnosis using the DSM.

A representative sample of geriatric patients for whom a delirium is suspected, will be recruited in the various participating centers, patients will undergo two consecutive visits:

* A visit by a geriatrician, during which the confused state of the patient will be evaluated using the French version of the CAM.
* A visit by a psychiatrist during which the diagnosis of confusional state will be evaluated using the gold standard criteria of the DSM IV.

These two evaluations will be conducted on the same day and blinded from each other.

The order of these two procedures will be balanced within each center. This process will allow the calculation of diagnostic parameters of the CAM French version (validation competitive): sensitivity, specificity, positive and negative predictive values .

ELIGIBILITY:
Inclusion Criteria:

* A family member of the patient, or his/her "trusted person" must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* Hospitalization in geriatric short stay OR patient consulting at a geriatric assessment center / memory clinic OR geriatric day hospitalization
* Patients for whom a state of confusion is suspected during the pre-inclusion visit run-in based on the following criteria:
* Presence of a cognitive function disorder as defined by a score greater than or equal to 3 on the Short Portable Mental Status Questionnaire (SPMSQ) (Pfeiffer E, 1975) AND / OR
* Presence of a mood disorder and / or behavior disorder (regardless of duration) according to the patient's family or caregivers
* Presence of a caregiver who can answer questionnaires concerning activities of everyday life

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient's family or "trusted-person" refuses to sign the consent
* The patient does not understand french
* Severe aphasia
* Stay is < = 3 days

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients 75 years or older for whom a state of confusion is suspected during hospitalization or during a consultation for a geriatric or memory assessment.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2014-04; Primary Completion 2016-02-11 (Actual); Study Completion 2016-02-11 (Actual)

PRIMARY OUTCOMES:
CAM French Version: diagnostic properties | Day 0
  Sensitivity, specificity, positive predictive value, negative predictive value

SECONDARY OUTCOMES:
Reliability and quality of the french version of the CAM | Day 0
  Parameters of reliability and quality of the tool:
  * Inter-rater Agreement (measured by a coefficient of correlation) between two evaluators: geriatrician and a nurse or psychologist
  * Internal consistency of the questionnaire assessed by calculating Cronbach's alpha
  * Time required for assessment
  * Acceptability by clinicians
  * Tolerance of patients
Feasibility of scoring with the French version of the Delirium Index | day 0
Diagnostic properties of alternative algorithms constructed from items of CAM (French version) | day 0

OTHER OUTCOMES:
Patient age (years) | Baseline (day 0)
Patient weight (kg) | Baseline (Day 0)
Height (cm) | Baseline (day 0)
Education level | baseline (day 0)
  primary, secondary, or higher
Living situation (qualitative) | baseline (day 0)
  Does the patient live at home? or is the patient institutionalized?
Presence/absence of a caregiver | baseline (day 0)
Hospitalization within the past 3 months? yes/no | baseline (day 0)
Has the patient fallen within the past year? yes/no | baseline (day 0)
presence/absence of a visual or hearing impairment | baseline (day 0)
patient position during evaluation | baseline (day 0)
  qualitative variable: in bed, in a wheelchair, sitting down
ADL (Activities of Daily Living) score for the 15 days preceding inclusion | baseline (day 0)
IADL (Instrumental Activities of Daily Living) score for the 15 days preceding inclusion | baseline (day 0)
ADL (Activities of Daily Living) score at the moment of inclusion | baseline (day 0)
Clinical and para-clinical examination | baseline (day 0)
Evaluation of the patient's physiological state | baseline (day 0)
Diagnosis | baseline (day 0)
Prescribed drugs | baseline (day 0)
Comorbidities (Charlson score) | baseline (day 0)
History of dementia, depression or another psychiatric disorder | baseline (day 0)
  Notification in the patient's history of dementia, depression or another psychiatric disorder, assessed by NPI-R and Mini GDS.
Severity of clinical condition | baseline (day 0)
  Severity of clinical condition: MEWS (Subbe CP et al, 2001) and CGI (Guy W 1976) + Charlson scale
Presence or absence of dementia before admission | baseline (day 0)
  Presence or absence of dementia before admission (IQCODE French version) (Jorm AF 1994 and Law S, 1995)

CONTACTS AND LOCATIONS:
Overall Officials: Valéry Antoine, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (8):
- France (8):
  - CH d'Alès, Alès
  - CHU de Rouen - Hôpital de Bois-Guillaume, Bois-Guillaume
  - APHP - Hôpital Charles Foix, Ivry-sur-Seine
  - APHM - Hôpital Sainte-Marguerite, Marseille
  - CHU de Montpellier - Centre Antonin Balmes, Montpellier
  - CHU de Nice - Hôpital de Cimiez, Nice
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - CHU de Reims - Hôpital Maison Blanche, Reims

REFERENCES:
- [Result] Antoine V, Belmin J, Blain H, Bonin-Guillaume S, Goldsmith L, Guerin O, Kergoat MJ, Landais P, Mahmoudi R, Morais JA, Rataboul P, Saber A, Sirvain S, Wolfklein G, de Wazieres B. [The Confusion Assessment Method: Transcultural adaptation of a French version]. Rev Epidemiol Sante Publique. 2018 May;66(3):187-194. doi: 10.1016/j.respe.2018.01.133. Epub 2018 Apr 4. French. PMID 29625860